CLINICAL TRIAL: NCT04358016
Title: The Protection of Telipression on Developing of Acute Kidney Injury in Cirrhotic Patients With Upper-gastroentestinal Bleeding
Brief Title: Terlipression Prevent Developing of Acute Kidney Injury During Upper-gastroentestinal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, LiangXS, Professor, Changhai Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LDWJPMF-102-1700
Record Dates: First submitted 2019-10-15; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2019-11

CONDITIONS: Cirrhosis, Liver; Upper Gastrointestinal Bleeding
Keywords: liver cirrhosis; upper gastrointestinal bleeding; acute kidney injury; urinary IL-18
MeSH Terms: conditions — Liver Cirrhosis; Gastrointestinal Hemorrhage; Acute Kidney Injury | interventions — Terlipressin; Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- terlipression (Experimental): terlipression 1mg；once every 6 hours；5days
  Interventions: Drug: Terlipressin
- Control (Active Comparator): Somatostatin，3mg， once every 12 hours; 5 days
  Interventions: Drug: Somatostatin

INTERVENTIONS:
Drug: Terlipressin — Evaluate the effect of Terlipression on the occurance of acute kidney injury in patients with upper-gastroentestinal bleeding
  Arms: terlipression
Drug: Somatostatin — Somatostatin
  Arms: Control

SUMMARY:
The investigators studied the renal function index level in terlipressin treated cirrhotic patients with upper-gastrointestinal bleeding at different time point.

DETAILED DESCRIPTION:
54 cirrhotic patients with uppre-gastrointestinal bleeding were entrolled and were distributed into terlipressin group and control group at 1:1 rate. Patients in Terlipressin group received 1mg/6h of terlipressin intravenously for 5 days, and patients in control group recerved 1mg/12h of Somatostatin intravenously for 5 days.

At enrollment, 24h,48h,72,and 1week, the renal function index level( serum creatinine,urine biochemistry and Urinary tubule injury index etc) were tested.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosied as cirrhosis with upper gastrointestinal bleeding 18≤age≤70 Varicose vein rupture occurred within 24 hours, Without drug, endoscopy or interventional therapy Can read, understand and sign informed consent

Exclusion Criteria:

* Pregnant women, lactating women; Serious cardiovascular disease: history of acute cardiac infarction, heart block, heart failure, arterial hypertension(（SBP>170mmHg and/ or DBP>100mmHg） Occlusive lower extremity venous disease Asthma, chronic obstructive pulmonary disease Have serious or unable to control other organ diseases; Cerebrovascular disease; Age ≥70 years old Known to be allergic to therapeutic drugs Chronic kidney disease Weight ≤40kg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
incidence of acute kidney injure | 48 hours
  serum creatinine level increased by 26.5umol/L during 48hours or increased 50% compared to baseline

SECONDARY OUTCOMES:
hemostasis rate | 48 hours
  Fecal occult blood negative or hemoglobin stable after 48H treatment
incidence of hepatic encephalopathy | 48 hours
  Increased blood ammonia or directional force and computational power decrease after 48H treatment
The incidence of spontaneous bacterial peritonitis; | 48 hours
  After 48H treatment, there is ascites and ascites has more than 20% nuclear cells
The incidence of hyponatremia | 48 hours
  Serum sodium levels below 130mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Xuesong Liang, Dr, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Changhai hospital, Shanghai, China